CLINICAL TRIAL: NCT01315496
Title: A Placebo-controlled, Randomized, Double-blind, Multi-center, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous Administration of 'IV-Globulin S Inj.' in Adult Subjects With Community-Acquired Severe Sepsis or Septic Shock
Brief Title: GCIV as an Adjuvant Therapy for Community-Acquired Severe Sepsis or Septic Shock
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCIV_P3
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Human Immunoglobulin G; Sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Immunoglobulin G

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imunoglobulin G (Experimental): The enrolled patients will be randomized to receive supplementation of IVIG in ICU within 48 hours after hospital arrival admission for 3 consecutive days.
  Interventions: Drug: Immunoglobulin G
- Placebo control (Placebo Comparator): The enrolled patients will be randomized to receive supplementation of placebo (0.9% NaCl) in ICU within 48 hours after hospital arrival admission for 3 consecutive days.
  Interventions: Drug: Immunoglobulin G

INTERVENTIONS:
Drug: Immunoglobulin G — Immunoglobulin 1.5-2g/Kg/3days
  Other Names: GCIV

SUMMARY:
This study is to determine whether the intravenous application of 'Ⅳ-Globulin S inj. (Human Immunoglobulin G)' can reduce mortality in patients with severe sepsis or septic shock.

DETAILED DESCRIPTION:
A Placebo-controlled, Randomized, Double-blind, Multi-center, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous Administration of 'IV-Globulin S inj.(Human Immunoglobulin G)' as an Adjuvant Therapy in Adult Subjects with Community-Acquired Severe Sepsis or Septic Shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis or septic shock, if all of the following criteria is satisfied.

  1. Age ≥ 18 years
  2. Proved or suspected infection in at least one site
* pneumonia
* urinary tract infection
* intra-abdominal infection
* primary bloodstream infection
* skin and soft tissue infection 3. Three or more of the following
* a core temperature ≥ 38° C or ≤ 36° C
* a heart rate ≥ 90 beats/min
* a respiratory rate ≥ 20 breaths/min or PaCO2 ≤ 32 mmHg or use of mechanical ventilation for an acute process
* a white blood cell count ≥ 12000/mm3 or ≤ 4000/ mm3 or immature neutrophils > 10% 4. Acute organ failure in one or more of the following
* kidney
* respiratory system
* blood system
* metabolic system
* circulatory system 5. APACHE score ≥ 20 and ≤ 29 6. Patient can treatment with GCIV in ICU within at least 48 hours 7. Informed consent

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. a weight > 100kg
3. discharged from the hospital at least 14 days prior to new admission
4. Transferred from another hospital staying more than 48 hours
5. allergy or shock of IVIG
6. Treated with IVIG within the 12 weeks immediately preceding enrolment in this study
7. IgA deficiency
8. Hypernatremia or hyperhydration
9. Proved or suspected HIV or AIDS patients(CD4+ <200mL)
10. Current participation in any study within the last 4 weeks
11. Do not resuscitate (DNR) status
12. Patient's death is considered imminent due to coexisting disease
13. physicians decision to exclude patients from this protocol
14. Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 28th day

SECONDARY OUTCOMES:
All cause mortality | 7th day
Course of SOFA subscores | 5 Times: D-1, D1, D3, D5, D7
Laboratory Test | 7th Day
  sputum culture test, CBC, blood chemistry, blood coagulation test, CRP, ABGA
Duration of ICU and general ward admission | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Min Ja Kim, Professor, Principal Investigator — Korea University Anam Hospital
Locations (17):
- South Korea (17):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Hospital, Incheon
  - Gyrongsang National University Hospital, Jinju-si, Gyeongsangnam-do,
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic of Korea Yeouido ST. Mary's Hospital, Seoul
  - Ajuo University Hospital, Suwon
  - Wonju Christian Hospital, Wŏnju